CLINICAL TRIAL: NCT03746275
Title: Xarelto + Acetylsalicylic Acid: Treatment Patterns and Outcomes in Patients With Atherosclerosis. A Non-interventional Study
Brief Title: Study to Gain Insights in Treatment Patterns and Outcomes in Patients With Atherosclerosis Prescribed to Xarelto in Combination With Acetylsalicylic Acid
Acronym: XATOA
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen, LP (Industry)
Responsible Party: Sponsor
Other Study IDs: 20280
Record Dates: First submitted 2018-11-01; First posted 2018-11-19 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Atherosclerosis
Keywords: Coronary artery disease (CAD); Peripheral artery disease (PAD); Major adverse limb events (MALE); Major adverse cardiac events (MACE); Atherosclerosis; Atherothrombosis; Thrombosis; Embolism; Thromboembolism
MeSH Terms: conditions — Atherosclerosis; Coronary Artery Disease; Peripheral Arterial Disease; Cardiovascular Diseases; Thrombosis; Embolism; Thromboembolism | interventions — Rivaroxaban; Aspirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CAD/PAD-patients: Adult patients with coronary artery disease (CAD) or symptomatic peripheral artery disease (PAD) from Europe, Asia, Latin America and Canada, who are treated with a combination of rivaroxaban and acetylsalicylic acid to prevent atherothrombotic events
  Interventions: Drug: Rivaroxaban (BAY59-7939, Xarelto); Drug: Acetylsalicylic acid

INTERVENTIONS:
Drug: Rivaroxaban (BAY59-7939, Xarelto) — 2.5 mg twice daily
  Other Names: Xarelto
Drug: Acetylsalicylic acid — 75 - 100 mg once daily according to local label
  Other Names: Aspirin

SUMMARY:
In this study researchers want to gain more information on treatment patterns of patients treated with Xarelto in combination with acetylsalicylic acid (ASA). Both drugs reduce the risk of blood clots via different pathways. The study will enroll adult patients suffering from coronary artery disease (narrowing or blockage of vessels that supply the heart with blood) or peripheral artery disease (narrowing or blockage of vessels that supply the legs or head with blood). The study will focus on information on when and why physicians are starting to treat patients with Xarelto in addition to ASA, treatment duration, reasons to discontinue treatment and previous therapies. The study will also look into treatment outcomes for patients being treated with a combination of Xarelto and ASA by their physicians.

DETAILED DESCRIPTION:
The study aims to collect real-world data on treatment patterns and decision points for treatment in patients with coronary artery disease (CAD) and/ or peripheral artery disease (PAD) treated with rivaroxaban 2.5 mg [twice daily] for the prevention of major cardiovascular events in adult patients with CAD at high risk of ischemic events and/ or documented PAD and to describe outcomes of an antithrombotic regime based on dual pathway inhibition (vascular dose of rivaroxaban 2.5 mg [twice daily] plus low-dose ASA [once daily]) across the broad range of patient risk profiles encountered in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Adults with diagnosis Coronary Artery Disease (CAD) or Peripheral Artery Disease (PAD).
* Treatment according to local marketing authorization, rivaroxaban 2.5 mg twice daily started within 4 weeks prior to enrolment. Only in those countries with a marketing authorization of rivaroxaban in the acute coronary syndrome (ACS) indication, also patients already on rivaroxaban treatment for ACS, who are subsequently fulfilling criteria for CAD, are allowed to be enrolled within 4 weeks of this decision being made.

Exclusion Criteria:

* Patients who will be treated with chronic anticoagulation therapy other than rivaroxaban 2.5 mg given for CAD/PAD.
* Participation in an interventional trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults in routine medical practice, multi-national
Sampling Method: Non-Probability Sample
Enrollment: 5798 (Actual)
Dates: Start 2018-11-13 (Actual); Primary Completion 2021-06-08 (Actual); Study Completion 2021-07-13 (Actual)

PRIMARY OUTCOMES:
Descriptive analysis of patient history of CAD | At baseline
Descriptive analysis of patient history of PAD | At baseline
Descriptive analysis of prior antithrombotic treatment | At baseline
Descriptive analysis of concomitant antithrombotic treatment | Up to 30.5 months
Descriptive analysis of prior secondary prevention therapies | At baseline
Descriptive analysis of concomitant secondary prevention therapies | Up to 30.5 months
Reason for start of rivaroxaban | At baseline
  Reasons include past ischemic events, co-morbidities and medical history.
Decision point for start of rivaroxaban | At baseline
  Time point of start of medication in relation to disease progress and/ or occurrence of ischemic events.
Reason for discontinuation of rivaroxaban | Up to 30.5 months
Planned duration of treatment with rivaroxaban | At baseline
Actual duration of treatment with rivaroxaban | Up to 30.5 months
Planned duration of treatment with acetylsalicylic acid | At baseline
Actual duration of treatment with acetylsalicylic acid | Up to 30.5 months

SECONDARY OUTCOMES:
Occurrence of major adverse cardiac events | Up to 30.5 months
  Composite measure of stroke, myocardial infarction and cardiovascular death
Occurrence of stroke | Up to 30.5 months
Occurrence of myocardial infarction | Up to 30.5 months
Occurrence of cardiovascular death | Up to 30.5 months
Occurrence of major adverse limb events | Up to 30.5 months
  Major adverse limb events comprise acute/severe limb ischemia including major amputation and chronic limb ischemia.
Occurrence of acute/severe limb ischemia | Up to 30.5 months
Occurrence of chronic limb ischemia | Up to 30.5 months
Occurrence of major amputation | Up to 30.5 months
Anti-thrombotic treatment pattern after major adverse limb event | Up to 30.5 months
  Treatment pattern comprises drug name, dose and duration of treatment.
Occurrence of thromboembolic events | Up to 30.5 months
  Thromboembolic events include systemic embolism and venous thromboembolism.
Occurrence of haemorrhagic events | Up to 30.5 months
  A haemorrhagic event is any event related to bleeding.
Occurrence of death from cardiovascular events | Up to 30.5 months
Occurrence of death from any cause | Up to 30.5 months
Occurrence of cardiac revascularization procedures | Up to 30.5 months
  Includes percutaneous coronary intervention and coronary artery bypass grafting.
Occurrence of peripheral revascularization procedures | Up to 30.5 months
Occurrence of carotid revascularization procedures | Up to 30.5 months
Occurrence of hospitalizations | Up to 30.5 months
  Hospitalizations due to stroke, cardiovascular reasons, major adverse limb events or bleeding complications.
Duration of hospitalization | Up to 30.5 months
  Time in days of hospitalization due to stroke, cardiovascular reasons, major adverse limb events or bleeding complications.
Total walking distance of PAD patients | Up to 30.5 months
Pain-free walking distance of PAD patients | Up to 30.5 months

CONTACTS AND LOCATIONS:
Locations (18):
- Multiple facilities, Multiple Locations, Argentina
- Multiple facilities, Multiple Locations, Brazil
- Multiple facilities, Multiple Locations, Canada
- Multiple facilities, Multiple Locations, Denmark
- Multiple facilities, Multiple Locations, Germany
- Multiple facilities, Multiple Locations, Israel
- Multiple facilities, Multiple Locations, Lebanon
- Multiple facilities, Multiple Locations, Luxembourg
- Multiple facilities, Multiple Locations, Mexico
- Multiple facilities, Multiple Locations, Norway
- Multiple facilities, Multiple Locations, Russia
- Multiple facilities, Multiple Locations, Slovenia
- Multiple facilities, Multiple Locations, South Korea
- Multiple facilities, Multiple Locations, Sweden
- Multiple facilities, Multiple Locations, Switzerland
- Multiple facilities, Multiple Locations, Thailand
- Multiple facilities, Multiple Locations, United Arab Emirates
- Multiple facilities, Multiple Locations, United Kingdom

REFERENCES:
- [Derived] Fox KAA, Anand SS, Aboyans V, Cowie MR, Debus ES, Zeymer U, Monje D, Vogtlander K, Lawatscheck R, Gay A. Xarelto plus Acetylsalicylic acid: Treatment patterns and Outcomes in patients with Atherosclerosis (XATOA): Rationale and design of a prospective registry study to assess rivaroxaban 2.5 mg twice daily plus aspirin for prevention of atherothrombotic events in coronary artery disease, peripheral artery disease, or both. Am Heart J. 2020 Apr;222:166-173. doi: 10.1016/j.ahj.2020.01.015. Epub 2020 Jan 28. PMID 32092505
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/